CLINICAL TRIAL: NCT05782712
Title: Rapid Measurement of Adenosine Concentration in Patients With Syncope
Brief Title: Rapid Measurement of Adenosine in Syncope Patients
Acronym: BlotSpot
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C130
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Syncope
Keywords: Syncope; Adenosine
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Syncope: patients referred for syncope evaluation
  Interventions: Biological: adenosine dosage
- No syncope: Subjects without syncope
  Interventions: Biological: adenosine dosage

INTERVENTIONS:
Biological: adenosine dosage — Whole blood is collected using finger puncture followed by deposit a drop of blood (20 μL) using finnpipette, on a blotting paper (Whatman 903 protein saver cards™) and dried over night at room temperature to obtain dried blood spot (DBS).

SUMMARY:
Until now, a barrier to the widespread evaluation of adenosine in clinical practice has been the difficulty of obtaining rapid reliable measures. A rapid method has recently been developed which consists of measuring adenosine concentration in whole blood instead of plasma by means of Mass Spectrometry (LC-MS/MS). In this study adenosine plasma levels were assessed in a larger unselected cohort of patients affected by non-cardiac syncope and compared the results with healthy controls.

DETAILED DESCRIPTION:
Rationale and aim Until now, a barrier to the widespread evaluation of adenosine in clinical practice has been the difficulty of obtaining rapid reliable measures. Indeed, owing to its short half-life in the blood, adenosine is not easy to sample and measure. At the time of venepuncture, a stop solution - not commercially available - must be utilized in order to inhibit the degradation of adenosine in body fluid. After plasma deproteinization, adenosine concentration is evaluated by means of high-performance liquid chromatography.

A rapid method has recently been developed which consists of measuring adenosine concentration in whole blood instead of plasma by means of Mass Spectrometry (LC-MS/MS). In brief, whole blood is collected after finger puncture and a drop is deposited on a blot paper (Whatman). After the extraction of adenosine by means of a mixture consisting of methanol and internal standard, its concentration is measured by LC-MS/MS. This method is rapid, well accepted by the patient, not expensive, and easily replicable. Comparison between the two above-mentioned methods in 20 healthy subjects and in patients with vasovagal syncope has shown an acceptable correlation, with a r=0.65 and p<0.01. The mean adenosine concentration was significantly higher in vasovagal syncope patients than in controls (3.1 µM versus 0.60 µM, p<0.001). However, the above results need to be replicated in a larger sample of patients and controls before the blot paper method of measurement of adenosine can replace the standard method.

In this study denosine plasma levels was assessed in a larger unselected cohort of patients affected by non-cardiac syncope and compared the results with healthy controls.

Study design The rapid method of adenosine dosage in whole blood was assessed in patients with syncope and in controls. The study was performed in patients referred to Istituto Auxologico Italiano. The blood sample was be shipped to the Laboratory of Biochemistry, Timone Hospital 264 Rue Saint-Pierre, 13385 Marseille, France for analysis Syncope group: patients referred to the Syncope Unit of Auxologico with a diagnosis of possible or certain reflex syncope (class I diagnostic criteria of ESC guidelines) after exclusion of competing diagnoses.

There syncope patients are subdivided in 3 predefined subgroups:

* Subgroup A) Patients with no prodromes or very short prodromes (5 sec), normal heart and normal ECG
* Subgroup B) Patients with typical vasovagal features (orthostatic or emotional triggers, long prodromes with signs and symptoms of autonomic activation, i.e, nausea, sweating, dizziness, pallor)
* Subgroup C) Patients who do not belong to none of the above subgroups.

No syncope group: 1) Patients without a history of syncope, referred to Auxologico for other reasons; these patients have absence of severe structural heart disease and other comorbidities. 2) Healthy volunteers selected among personnel of Auxologico. The selection of these patients will be made matching them to syncope cases by age and sex.

Blood samples collection Whole blood is collected using finger puncture followed by deposit a drop of blood (20 μL) using finnpipette, on a blotting paper (Whatman 903 protein saver cards™) and dried over night at room temperature to obtain dried blood spot (DBS).

Blood samples extraction Six millimeters of dried blood spot (DBS) are cut out followed by extraction with mixture consisting of methanol (400 μl) and internal standard (50 μl) in 2 mL microfuge tubes then mixed for 90 min at 45°C. After extraction, an aliquot of 350 μL are transferred into a new 2-mL safe-lock tube and evaporated to dryness at 60°C under nitrogen, 150 μl of 0.1% formic acid in water are added and quickly vortexed before transferring into an HPLC auto sampler vial.

Adenosine dosage After the extraction of adenosine by means of a mixture consisting of methanol and internal standard, its concentration is measured by LC-MS/MS.

Samples are analyzed using a Shimadzu UFLC XR system consisting of two LC-20ADXR binary pumps, a DGU-20A5R vacuum degasser, and a CT0-20AC thermostated column oven and a SIL-20ACXR cooled auto sampler (Shimadzu, Marne la Vallee, France). The LC system was interfaced with an ABSciex 4500 triple quadrupole mass spectrometer (Les Ulis, France) operating with an electrospray ionization source (ESI) using nitrogen (purity: 99.99%). Ten microliters of the extracted sample were injected onto a 2.1 × 100 mm, 3 μm AtlantisR T3 column, Waters (Guyancourt, France). The starting mobile phase consisted of 3% methanol and 97% acidified water (0.1% formic acid) with a flow of 0.7 ml/min for 3.5 min. Then, the gradient of methanol was increased to 30% for 3 min. The column was re- equilibrated for 2 min to starting conditions.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the Syncope Unit of Auxologico with a diagnosis of possible or certain reflex syncope (class I diagnostic criteria of ESC guidelines)

Exclusion Criteria:

* exclusion of competing diagnoses.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Syncope group: patients referred to the Syncope Unit of Auxologico with a diagnosis of possible or certain reflex syncope (class I diagnostic criteria of ESC guidelines) after exclusion of competing diagnoses.
  No syncope group: 1) Patients without a history of syncope, referred to Auxologico for other reasons; these patients have absence of severe structural heart disease and other comorbidities. 2) Healthy volunteers selected among personnel of Auxologico. The selection of these patients will be made matching them to syncope cases by age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Adenosine dosage | 2 hours
  Comparison of plasmatic adenosine value observed in the syncope group with that of control group

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: Upon reasonable request after the publication of the principal study
Access Criteria: m.brignole@auxologico.it